CLINICAL TRIAL: NCT05996328
Title: CSP #2025 - Geriatric OUt-of-hospital Randomized MEal Trial in Heart Failure: Veterans Affairs (GOURMET-VA)
Acronym: GOURMET-VA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Two-arm study: active intervention vs study-defined standard of care
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants, dietitians, and site coordinators can't be blinded. However, the investigators and outcome assessors will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Study-defined standard of care
  Interventions: Other: Study -defined standard of care
- Home-delivered meals and short-term dietary counseling (Experimental): Home-delivered, low-sodium, nutritionally robust meals for 6 weeks plus two additional remotely delivered dietary counseling sessions in addition to the study-defined standard of care.
  Interventions: Other: Home-delivered meals and short-term dietary counseling

INTERVENTIONS:
Other: Home-delivered meals and short-term dietary counseling — Home-delivered, low-sodium, nutritionally robust meals for 6 weeks plus two additional remotely delivered dietary counseling sessions in addition to the study-defined standard of care.
  Arms: Home-delivered meals and short-term dietary counseling
Other: Study -defined standard of care — study-defined standard of care consists of standardized dietary education and a single dietary counseling session shortly after discharge
  Arms: Control

SUMMARY:
The purpose of this multi-center clinical trial is to study the efficacy and safety of providing nutritional support added to the study-defined standard of care which consists of standardized dietary education and a single dietary counseling session shortly after discharge, versus study-defined standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years
* Veterans enrolled in a VHA facility
* Hospitalized ( 24 hours) with new HF or worsening chronic HF
* Dentition, swallowing function, etc. sufficient to safely consume food and liquid of standard composition and texture (i.e., no pureed food, no thickened liquids needed)
* Able and willing to provide informed consent and perform study activities

Exclusion Criteria:

* Food allergies or intolerances that cannot be accommodated by study diet
* On dialysis or estimated glomerular filtration rate <30 at randomization
* Serum potassium (non-hemolyzed) >6.0 mmol/L during index hospitalization
* Heart transplant or active transplant listing
* Left ventricular assist device present or anticipated <6 months
* Malignancy or other non-cardiac condition limiting life expectancy to <12 months
* Planned admission to a skilled nursing facility following hospital discharge, or discharge to other location/situation where Veteran does not have control over diet
* Lack of space to store food for a week or equipment to prepare food
* Severe cognitive impairment (SLUMS score <20, or <19 if less than high school education completed)
* Severe food insecurity (5 or 6 points on the USDA 6-item Food Insecurity Screen)
* Body mass index >50 kg/m2
* Other medical, psychiatric, behavioral, or logistical condition which, in the clinical judgement of the site investigator, makes it unlikely the patient can effectively participate in or complete the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of pairwise comparisons with wins of Clinical Benefit, evaluated a hierarchical composite of days alive out of hospital and =5-point difference in the change of health-related quality of life | within 6 weeks post-index hospital discharge
  All patients randomized to intervention are compared to all patients randomized to placebo within strata. In each comparison with any two patients, a patient will win by achieving a superior clinical outcome which is determined by sequentially assessing the following criteria with evaluation halted when distinct advantage for either patient is shown:
  1. Days alive out of hospital at 6 weeks: shorter days is worse; tied, if same days alive out of hospital. Move to evaluation of 2 if tied.
  2. Change of The Kansas City Cardiomyopathy Questionnaire Clinical Summary (KCCQ-CS) at 6 weeks from baseline: the threshold for the difference is greater or equal to 5 for a win; tied, if difference is less than 5.
  The KCCQ-CS ranges from 0 to 100, where a higher score reflects a better outcome.

SECONDARY OUTCOMES:
DAOH at 6 months post-discharge | 6 months post-discharge
  This outcome was selected to determine whether home-delivered meals, augmented by enhanced dietary counseling, during a high-risk period have durable effects on readmission burden.

CONTACTS AND LOCATIONS:
Overall Officials: Scott L. Hummel, MD, Study Chair — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Digital data underlying primary scientific publications from this study will be held as part of a data sharing resource maintained by the Cooperative Studies Program (VA-CSP). These data may be available to the public and other VA and non-VA researchers under certain conditions and consistent with the informed consent and CSP policy which prioritize protecting subjects' privacy and confidentiality to the fullest extent possible